CLINICAL TRIAL: NCT04835142
Title: Phase III Clinical Study Comparison of A140 and Erbitux Combined With mfolfox6 to Evaluate Efficacy and Safety of First-line Treatment for Ras Wild-type mCRC
Brief Title: Comparison of A140 and Erbitux Combined With mfolfox6 to Evaluate Efficacy and Safety of First-line Treatment for Ras Wild-type mCRC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KL140-Ⅲ-02-CTP
Record Dates: First submitted 2021-03-15; First posted 2021-04-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: RAS wild-type; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double blind control period (Experimental): experiment arm： All eligible subjects will receive A140 in combination with mFOLFOX-6 chemotherapy regimen every 2 weeks.
  control arm: All eligible subjects will receive Erbitux in combination with mFOLFOX-6 chemotherapy regimen every 2 weeks.
  Interventions: Drug: Double blind control period A140
- Open single period (Experimental): All eligible subjects will receive A140 in combination with mFOLFOX-6 chemotherapy regimen every 2 weeks.
  Interventions: Drug: Open single period A140

INTERVENTIONS:
Drug: Double blind control period A140 — experiment arm： Drug A140:400 mg/m2（D1，iv）,250 mg/m2（qw，iv） Drug Oxaliplatin 85 mg/m2（D1,iv), Drug Calcium Folinate 400 mg/m2（D1,iv） Drug 5-FU 400 mg/m2（D1,iv），2400 mg/m2 (48±4h) control arm: Drug Erbitux:400 mg/m2（D1，iv）,250 mg/m2（qw，iv） Drug Oxaliplatin 85 mg/m2（D1,iv) Drug Calcium Folinate 400 mg/m2（D1,iv） Drug 5-FU 400 mg/m2（D1,iv），2400 mg/m2 (48±4h)
  Other Names: KL-140
  Arms: Double blind control period
Drug: Open single period A140 — Drug A140:400 mg/m2（D1，iv）,250 mg/m2（qw，iv） Drug Oxaliplatin 85 mg/m2（D1,iv), Drug Calcium Folinate 400 mg/m2（D1,iv） Drug 5-FU 400 mg/m2（D1,iv），2400 mg/m2 (48±4h)
  Other Names: KL-140
  Arms: Open single period

SUMMARY:
Compare the objective remission rate of A140 and Erbitux combined with mfolfox6 regimen in the first-line treatment of Ras wild-type metastatic colorectal cancer for 12 weeks

DETAILED DESCRIPTION:
In this study, a multicenter, randomized, double-blind, controlled trial design was used to compare the efficacy and safety of A140 or Erbitux combined with mfolfox6 regimen in the first-line treatment of Ras wild-type metastatic colorectal cancer patients

Objective to compare the 12 week objective response rate (ORR) of A140 and ebitur combined with mfolfox6 regimen in the first-line treatment of Ras wild-type metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Be able to understand the procedures and methods of this study, be willing to strictly abide by the clinical trial protocol to complete this trial, and sign the informed consent voluntarily
* Male or female subjects aged 18-75 years (including 18 and 75 years)
* Histologically proven diagnosis of metastatic colorectal cancer. No previous systemic chemotherapy for metastatic colorectal cancer. Patients who have completed adjuvant chemotherapy before the start of the study can be enrolled, Platinum containing chemotherapy needs to end for more than 12 months, and non platinum containing chemotherapy needs to end for more than 6 months;
* KRAS and NRAS genotypes in tumor tissues were wild type, and BRAF-V600E mutation was not found；
* At least one measurable lesion by computer tomography(CT) or magnetic resonance imaging (MRI)according to RECIST1.1 criteria (not in an irradiated area)
* Eastern Cooperative Oncology Group(ECOG)performance status of 0 or 1 at trial entry；
* Life expectancy of at least 16 weeks；
* The level of organ function before the first medication met the following requirements:

  1. Peripheral blood cell count: leukocyte count ≥ 3×10ˆ9 / L, neutrophil count ≥ 1.5× 10ˆ9 / L, platelet count ≥ 75 × 10ˆ9 / L, hemoglobin ≥ 90 g / L;
  2. Liver function: total bilirubin ≤ 1.5 ULN, Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 ULN; AST and ALT≤ 5 ULN in subjects with liver metastasis;
  3. Renal function: serum creatinine ≤ 1.5 ULN.
* Fertile subjects (male and female) were required to receive effective medical contraceptive measures until 3 months after the last study (see Annex 4 for specific contraceptive measures).

Exclusion Criteria:

* Those who are known to have an allergic reaction to any component of the study drug；
* Local treatments such as radiotherapy, radiofrequency ablation, intervention, etc or surgical procedures (excluding prior diagnostic biopsy) in the 28 days before first administration；
* Known brain metastasis and/or leptomeningeal disease；
* People with complete intestinal obstruction and incomplete intestinal obstruction requiring treatment. However, patients whose obstruction is relieved by fistula or stent placement can be included in the group;
* Active severe clinical infection (> Grade 2, NCI-CTCAE version 5.0), including active tuberculosis；
* Uncontrolled diabetes (fasting blood glucose ≥10 mmol/L), severe lung disease (such as acute lung disease, pulmonary fibrosis that affects lung function, interstitial lung disease. Except for radiation pneumonia that has recovered), liver failure；
* Clinically significant cardiovascular diseases, such as heart failure (NYHAⅢ-Ⅳ), uncontrolled coronary heart disease, cardiomyopathy, arrhythmia, hypertension (systolic blood pressure>150mmHg and/or diastolic blood pressure>100mmHg), echocardiography The figure shows the ejection fraction <50%, the history of myocardial infarction within the past two years；
* Renal replacement therapy；
* > Grade 1 Peripheral Nerve Disorder (NCI-CTCAE Version 5.0)；
* History of organ allograft, autologous stem cell transplantation, or allogeneic stem cell transplantation；
* Previous malignancy other than CRC in the last 5 years except basal cell cancer of the skin or preinvasive cancer of the cervix；
* HIV infection, hepatitis B surface antigen positive (and peripheral blood hepatitis B virus deoxynucleotide HBV DNA ≥ 1×10ˆ4 copy number/ml or ≥ 2000 IU/ml), hepatitis C virus antibody positive (and peripheral blood hepatitis C virus nucleotide HCV RNA≥ 1×10ˆ3 copies/ml or ≥ 200 IU/ml)；
* Patients with coagulation dysfunction, meet any of the following conditions: prothrombin time (PT) ≥ 1.5 ULN， thrombin time (TT) ≥ 1.5 ULN,activated partial thromboplastin time (APTT) ≥ 1.5 ULN;
* Previously treatment with VEGF pathway targeted therapy and EGFR monoclonal antibody；
* Past treatment history:

  1. Receiving other anti-tumor treatments (including anti-tumor treatments with traditional Chinese medicines, such as Aidi injection, Kanglaite injection, Kangai injection, cininobufosin, brucea javanica oil, etc.) within 4 weeks before the first administration of the study ；
  2. Long-term systemic immunotherapy, or hormone therapy for anti-tumor purposes (physiological replacement therapy, except for those with hypothyroidism who take thyroxine);
  3. Have received G-CSF, GM-CSF, whole blood or blood component transfusions within 4 weeks before the first medication of the study;
  4. Have received other experimental drugs or interventional clinical studies within 4 weeks before the first medication of the study；
* Pregnancy (confirmed by blood pregnancy test) or lactation；
* There is currently alcohol or drug dependence；
* There is a clear neurological disease or mental illness that has not been cured, including epilepsy, dementia, schizophrenia, etc；
* Adverse events of previous treatment (except for hair loss) did not return to grade 1 or below (NCI-CTCAE version 5.0)；
* The researcher believes that the patient has other factors that affect the efficacy or safety evaluation of this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
ORR | 16 Weeks
  The objective tumor response rate (ORR) of colorectal cancer patients at 12 weeks based on the evaluation of the independent imaging evaluation committee, and confirmed at least 4 weeks later

SECONDARY OUTCOMES:
ORR | 16 Weeks
  1)Based on the researcher's assessment of the objective tumor response rate (ORR) of patients with colorectal cancer after 12 weeks of medication, and confirmed at least 4 weeks later
Progression-free survival (PFS) | PFS-1 year
  2)PFS within 1 year after medication based on the evaluation by the independent imaging evaluation committee and the investigator
Overall survival (OS) | OS-1year
  2) OS within 1 year after medication based on the evaluation by the independent imaging evaluation committee and the investigator
Progression-free survival (PFS) | PFS-1 year after the last patient's first dose
  3)Based on the researcher's assessment of PFS after 1 year of medication
Overall survival (OS) | OS-1 year after the last patient's first dose
  3)Based on the researcher's assessment of OS after 1 year of medication

CONTACTS AND LOCATIONS:
Locations (1):
- 307 Hospital of PLA, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu R, Yin X, Bai Y, Zhong H, Ye F, Wang Q, Liu M, Li N, Deng Y, Wang Y, Xu J, Li W, Chen K, Cai S, Yang J, Zhang T, Li Y, Qin B, Deng L, Liu S, Li S, Si J, Li Y, Ge J, Xu N, Xu J. A140 plus mFOLFOX6 compared with cetuximab plus mFOLFOX6 for first-line RAS wild-type metastatic colorectal cancer: A randomized clinical trial. Eur J Cancer. 2025 Aug 26;226:115566. doi: 10.1016/j.ejca.2025.115566. Epub 2025 Jun 7. PMID 40737898